CLINICAL TRIAL: NCT02624297
Title: Effect of Exercise Training on Chemoreflex Control of Sympathetic Activity in Patients With Coronary Artery Disease and Obstructive Sleep Apnea
Brief Title: Chemoreflex Control of Sympathetic Activity in Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAD-2015/01
Record Dates: First submitted 2014-03-24; First posted 2015-12-08 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease (CAD); Obstructive Sleep Apnea (OSA)
Keywords: Coronary artery disease; Chemoreceptors; Sympathetic nerve activity; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Sleep Apnea, Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control Group (No Intervention): Healthy control group for comparisons with coronary artery disease groups.
- CAD without OSA - Control (No Intervention): Clinical follow-up.
- CAD without OSA - Intervention (Experimental): Aerobic exercise training.
  Interventions: Other: Aerobic exercise training
- CAD with OSA - Control (No Intervention): Clinical follow-up.
- CAD with OSA - Intervention (Experimental): Aerobic exercise training.
  Interventions: Other: Aerobic exercise training

INTERVENTIONS:
Other: Aerobic exercise training — The patients will be submitted to four months of aerobic exercise training, three time a week.
  Arms: CAD with OSA - Intervention; CAD without OSA - Intervention

SUMMARY:
The investigators hypothesize that chemoreflex response of muscle sympathetic nerve activity (MSNA) during hypoxia and hypercapnia will be increased in coronary artery disease (CAD) patients and that the presence of obstructive sleep apnea (OSA) will potentiate these responses. And, that the exercise training would decrease the chemoreflex response of MSNA in these patients.

DETAILED DESCRIPTION:
Forty patients with coronary artery disease, with (n=20) and without (n=20) obstructive sleep apnea will be studied. A healthy control, age-paired group (n=10) will be also evaluated. The patients will be submitted to a polysomnography and randomized for clinical follow-up or exercise training for four months. It will evaluated the autonomic function, chemoreflex control of sympathetic activity during hypoxic and hypercapnic maneuvers, endothelial function and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable coronary artery disease; Age between 35-60 years, male and female; BMI <30 kg/m2 Not involved in a regular exercise program at least three months before the survey;

Exclusion Criteria:

* Patients with angina and / or ischemia,
* Patients with diabetic neuropathy and / or ischemia of the lower limbs;
* Previous diagnosis of chronic pulmonary, neurological and orthopedic diseases, neoplasia, renal failure and insulin-dependent diabetes mellitus;
* Patients with acute myocardial infarction, cardiac surgery or hospitalization of cardiac origin six months before the study and carriers of pacemaker / implantable defibrillator;
* Patients with cardiac dysfunction (ejection fraction of left ventricle <40%);
* Current smoking and pregnant women.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Chemoreflex control of MSNA at rest and during exercise. | baseline and after 4 months
  Chemoreflex control of MSNA will be measured by microneurography technique during the gas mixture known exposure at rest and during exercise

SECONDARY OUTCOMES:
Endothelial Function | baseline and after 4 months
  Endothelial Function will be measured by markers present in blood samples.
Neurovascular Control | baseline and after 4 months
  Neurovascular Control will be measured by venous occlusion plethysmography technique during the exposure mixture of gases known at rest and during exercise.
Inflammatory markers | baseline and after 4 months
  Inflammatory markers will be measured by markers present in blood samples.
Quality of Life | baseline and after 4 months
  Quality of life will be measured by the questionnaire Short-Form Health Survey (SF-36).
Anxiety Trait and State | baseline and after 4 months
  Anxiety Trait and State will be measured by the Spielberger state trait anxiety inventory (STAI).
Symptoms of Depression | baseline and after 4 months
  The level of symptoms of depression will be measured by the Beck scale.
Mood State | baseline and after 4 months
  Mood State will be measured by the profile of mood states (POMS) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Urbana PB Rondon, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute (InCor) - University of Sao Paulo, São Paulo, Brazil